CLINICAL TRIAL: NCT05433376
Title: Clinical Trial of the ShOckwave Coronary Intravascular Lithotripsy (IVL) System Used to Treat CalcIfied Coronary ArtEries (SOLSTICE)
Brief Title: SOLSTICE Trial in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genesis Medtech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-PI-CIP001
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Calcifications Vascular
MeSH Terms: conditions — Coronary Artery Disease; Vascular Calcification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVL group (Experimental)
  Interventions: Device: Shockwave Coronary Intravascular Lithotripsy (IVL) System C2

INTERVENTIONS:
Device: Shockwave Coronary Intravascular Lithotripsy (IVL) System C2 — lithotripsy-enabled, low-pressure dilatation balloon to modify severely calcified lesions

SUMMARY:
This is a small sample size clinical trial in Chinese population to assess the safety and effectiveness of the Shockwave Coronary Intravascular Lithotripsy (IVL) System to treat de novo, calcified, stenotic, coronary lesions prior to stenting.

ELIGIBILITY:
Inclusion Criteria:

General

1. Subject ≥18 and ≤80 years of age，male or female.
2. Subjects with native coronary artery disease (including stable or unstable angina and silent ischemia) suitable for PCI
3. Subject or legally authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures

   Angiographic
4. Evidence of calcification at the lesion site by, a) angiography, with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion, OR by b) OCT, with presence of ≥270 degrees of calcium on at least 1 cross section
5. The lesion length must not exceed 40 mm
6. The target vessel reference diameter must be ≥2.5 mm and ≤4.0 mm
7. de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches), per investigator's assessment with:

   1. Stenosis of ≥70% and <100% or
   2. Stenosis ≥50% and <70% (visually assessed) that is deemed qualified for PCI by investigator
8. The target vessel must have TIMI flow 3 at baseline (visually assessed; may be assessed after pre-dilatation)
9. Ability to pass a 0.014" guide wire across the lesion

Exclusion Criteria:

General

1. Any comorbidity or condition which may reduce compliance with this protocol, including follow-up visits
2. Subject experienced an acute MI (STEMI or non-STEMI) within 30 days prior to index procedure
3. Subjects with cardiogenic shock or acute left heart failure; New York Heart Association (NYHA) class III or IV heart failure; left ventricular ejection fraction (LVEF) ≤ 35% within 6 months prior to the procedure (Note: if multiple LVEF assessments were performed, the measurement closest to index procedure will be chosen; it can be assessed in the procedure);
4. History of a stroke or transient ischemic attack (TIA) within 6 months, or any prior intracranial hemorrhage or permanent neurologic deficit
5. Uncontrolled diabetes defined as a HbA1c ≥10%
6. Non-coronary interventional or surgical structural heart procedures (e.g., TAVR, MitraClip, LAA or PFO occlusion, etc.) within 30 days prior to the index procedure
7. Subject refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
8. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
9. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint
10. Subject is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment); Or plans to become pregnant within 13 months after the study procedure;
11. Unable to tolerate dual antiplatelet therapy (i.e., aspirin, and either clopidogrel, prasugrel, or ticagrelor) for at least 6 months (for patients not on oral anticoagulation)
12. Subject has an allergy to imaging contrast media which cannot be adequately pre-medicated
13. Renal failure with serum creatinine >2.5 mg/dL or chronic dialysis
14. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months
15. Untreated pre-procedural hemoglobin <10 g/dL or intention to refuse blood transfusions if one should become necessary
16. Coagulopathy, including but not limited to platelet count <100,000 or International Normalized ratio (INR) > 1.7 (INR is only required in subjects who have taken warfarin within 2 weeks of enrollment)
17. Subject has a hypercoagulable disorder such as polycythemia vera, platelet count >750,000 or other disorders
18. Biomarkers [troponin or CK-MB] greater than the upper laboratory normal limit within 72 hours prior to index procedure (note: if both biomarkers are available, both must be normal)
19. Subject has an active systemic infection on the day of the index procedure with either fever, leukocytosis or requiring intravenous antibiotics
20. Subjects with a life expectancy of less than 1 year
21. Planned use of atherectomy, laser or scoring or cutting balloon, or any investigational device other than lithotripsy Angiographic
22. Previous stent within the target vessel implanted within the last year
23. Previous stent within 10 mm of the target lesion regardless of the timing of its implantation
24. Angiographic evidence of a dissection (≥ grade C) in the target vessel at baseline or after guidewire passage
25. Lesions in non-target vessels requiring PCI as below should be excluded:

    1. 24 hours to 30 days prior to the study procedure if the procedure was unsuccessful or complicated; or
    2. In 24 hours prior to the study procedure
    3. >30 days after the study procedure
26. Non-target lesion is including left main lesion with diameter stenosis ≥30%
27. Target vessel is too tortuous to deliver a stent assessed by investigators.
28. Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel
29. Evidence of aneurysm in target vessel within 10 mm of the target lesion
30. Target lesion is an ostial location (LAD, LCX, or RCA, within 5 mm of ostium) or an unprotected left main lesion.
31. Target lesion is a bifurcation with ostial diameter stenosis ≥30%
32. Second lesion with >50% stenosis in the same target vessel as the target lesion including its side branches
33. Target lesion is located in a native vessel that can only be reached by going through a saphenous vein or arterial bypass graft
34. Other situations not suitable for enrollment assessed by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-11-26 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | in 24 hours post-procedure or prior to discharge, whichever comes first
  defined as stent delivery with a residual stenosis <50% (core laboratory assessed, angiographically) and without in-hospital MACE
Freedom from major adverse cardiac events (MACE) within 30 days of the index procedure. | 30 days post index procedure
  MACE is defined as:
  * Cardiac death; or
  * Myocardial Infarction (MI) defined as CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave at discharge (periprocedural MI) and using the Fourth Universal Definition of Myocardial Infarction beyond discharge (spontaneous MI); or
  * Target Vessel Revascularization (TVR) defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing
  - Beijing Friendship Hospital,Capital Medical University, Beijing
  - Chinese Peoples Liberation Army General Hospital, Beijing